CLINICAL TRIAL: NCT00783055
Title: Autonomy Among Physically Frail Older People in Nursing Homes: a Study Protocol for an Intervention Study
Brief Title: Autonomy Among Physically Frail Older People in Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Mette Andresen/Senior Lecturer & PhD student, The University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2004-1-52G
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2008-10-31 (Estimated); Status verified 2008-08

CONDITIONS: Frailty
Keywords: Autonomy; Older people; Physically frail; Nursing home; Intervention study
MeSH Terms: conditions — Frailty | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): 12 weeks of individually tailored intervention programmes based on participants individual wishes for daily activities e.g.ADL, mobility, social, mental or creative that they want to improve, conserve - and/or to revive.
  Interventions: Other: Individually tailored programmes

INTERVENTIONS:
Other: Individually tailored programmes — Individualised intervention programmes based on individual wishes for daily activities
  Other Names: activity; autonomy

SUMMARY:
The purpose of this study is to assess the status of perceived autonomy and to evaluate the effectiveness of individually tailored programmes on perceived autonomy in physically frail older people living in nursing homes.

DETAILED DESCRIPTION:
Experiencing autonomy is recognised to promote health and well-being for all age groups. Perceived lack of control has been found to be detrimental to physical and mental health. There is a lack of evidence-based knowledge elucidating how frail older people in nursing home settings perceive autonomy. Further, there are no studies on the extent to which this perception can be influenced positively by participating in an individually tailored programme based on individual wishes for daily activities.

The purpose of this study was to evaluate the effectiveness of individually tailored programmes on perceived autonomy in physically frail older people in nursing homes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older
* All kinds of diseases leading to physical frailty
* Dependent on assistance in minimum one P-ADL activity
* Able to understand verbal instructions
* Willing to participate
* Expected to live in the nursing home during the 24 weeks
* Both men and women

Exclusion Criteria:

* Terminal stages of disease
* MMSE-score below 16

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 66 (Actual)
Dates: Start 2005-03; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
The Autonomy Sub-dimension | baseline, after 12 weeks, anfter 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lis Puggaard, PhD, Study Director — University of Southern Denmark
Locations (1):
- Centre of Applied and Clinical Excercise Sciences, Institute of Sports Science and Clinical Biomechanics, University of Southern Denmark, Odense, Denmark

REFERENCES:
- [Derived] Andresen M, Puggaard L. Autonomy among physically frail older people in nursing home settings: a study protocol for an intervention study. BMC Geriatr. 2008 Dec 1;8:32. doi: 10.1186/1471-2318-8-32. PMID 19040767